CLINICAL TRIAL: NCT03813719
Title: Anxiety and Distress Levels in Women With Suspected Endometrial Cancer Seen in the Rapid Access Gynaecology Clinic
Brief Title: Anxiety and Distress Levels in Women With Suspected Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 16HH3687 Psych Study EC
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Endometrial Cancer; Cancer; Uterine Cancer; Anxiety; Stress; Psychological
Keywords: endometrial cancer; cancer; uterine cancer; anxiety; stress; psychological; survey; point-of-care
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Uterine Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients attending Rapid access Gynaecology Clinic: All patients attending Rapid access Gynaecology Clinic for the first time.

SUMMARY:
Patients attending the rapid access gynaecology clinic with a suspicion of endometrial cancer are understandably nervous. Few studies have quantified anxiety and distress of patients in this group.

This study surveys anxiety and stress levels of women attending clinic (by filling in an anonymous questionnaire). Additionally, in women who need a tissue biopsy, women are asked to rate their pain scores.

DETAILED DESCRIPTION:
Aims:

Quantify the anxiety and stress levels of women attending the Rapid access gynaecology clinic with a suspicion of cancer

Background:

Endometrial cancer is a tumour originating in the endometrium (womb lining); it is the most common gynaecological cancer in the United Kingdom (UK). In 2012, there were almost 100,000 new cases diagnosed in Europe. Endometrial cancer classically presents with postmenopausal bleeding (bleeding after the menopause), or intermenstrual bleeding (bleeding in between periods).

Although routine management for these women does vary, in general a screening test is performed, typically a pelvic (internal) ultrasound to assess the endometrium (womb lining). In cases where the endometrial thickness is above the threshold for investigation -an endometrial biopsy (sampling cells from the womb lining) is indicated. Whilst well tolerated, this can be quite painful.

Once the endometrial biopsy is performed, it is sent to the histologist for further examination. Histological analysis may take several days and patients are either brought back to clinic for discussion of the results or are given a telephone appointment. The patient often will not know the result of the test for up to 2 weeks; thus causing a lot of unnecessary anxiety and distress.

The study:

Patients attending the Rapid Access Gynaecology Clinic will be invited to participate in the study by filling in a short anonymous survey.

Additionally, patients undergoing a tissue biopsy sample will be asked to provide a pain score, followed by a brief interview to ascertain if they would undergo the procedure again if it was needed and how they tolerated the procedure. Additionally, the time taken to perform the procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting to rapid access gynaecology clinic with suspected gynaecological cancer

Exclusion Criteria:

* Anyone lacking capacity.
* <18years old.
* Pregnant.
* Anyone unable to understand English (in absence of translator)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study on suspected endometrial cancer
Study Population: All women attending Rapid access gynaecology clinic in imperial College NHS trust
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Charlotte and Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consective patients attending Rapid access Gynaecology Clinic for the first time, with suspected endometrial cancer between July 2018 and April 2019
Period: Overall Study
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
Started | 250
Completed | 250
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients recruited from 2 London hospitals
Groups:
- All Patients Attending Rapid Access Gynaecology Clinic: Consecutive patients attending Rapid access Gynaecology Clinic for the first time with suspected endometrial cancer.
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
Number analyzed (Participants) | 250
Age, Customized [Count of Participants; unit: Participants]
  <30 | 13
  30-39 | 15
  40-49 | 43
  50-59 | 88
  60-69 | 56
  70-79 | 25
  80+ | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Caucasian | 141
  Race/ethnicity: Black/Afro-carribean | 34
  Race/ethnicity: Asian | 35
  Race/ethnicity: Mixed | 5
  Race/ethnicity: Other | 33
  Race/ethnicity: Prefer not to say | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 250

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Score for Patients Attending Clinic
Description: GAD 7 score - (Generalised Anxiety Disorder assessment 7 score). 7 items each measured and score summated. Scale 0-21.Cut offs 0-5, 6-10, 11-15, 16+ correlate with anxiety score. Higher levels = worse anxiety
Time Frame: Immediately before clinic (waiting room)
Population: GAD 7 scores were calculated for each patient
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- All Patients Attending Rapid Access Gynaecology Clinic: All patients attending Rapid access Gynaecology Clinic for the first time with suspected endometrial cancer.
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
Number analyzed (Participants) | 250
score on a scale | 6 [3 to 12]

2. Secondary Outcome: Pain Score if Needing a Tissue Biopsy
Description: Patients asked to rank Pain score (using visual analogue score standardised tool), 0 to 10 score, where 0 is no pain and 10 is the worst pain in their life.
Time Frame: Immediately after tissue sample taken.
Population: Only 23 women required a tissue biopsy
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
Number analyzed (Participants) | 23
score on a scale | 5.5 [3 to 8]

3. Secondary Outcome: Time Taken for Tissue Sample to be Performed
Description: Measure time taken to perform tissue sample (in minutes) from insertion to removal of speculum.
Time Frame: During tissue biopsy time
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
Number analyzed (Participants) | 23
Minutes | 5.5 [3 to 8]

ADVERSE EVENTS:
Time Frame: Survey and paired observational study. No additional interventions performed (pipelle biopsies were part of standard of care) so adverse effects specifically due to study should be zero. Having said that, the time and pain score for pipelle biopsies were observed and recorded as part of this study and complications for pipelle biopsy were recorded. Any complications for a tissue biopsy would be apparent immediately, so time frame post biopsy 20 minutes.
Description: Survey and Observational study.
Arm/Group | All Patients Attending Rapid Access Gynaecology Clinic
All-Cause Mortality (participants affected / at risk) | 0/250
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT03813719/Prot_SAP_000.pdf